CLINICAL TRIAL: NCT05014256
Title: System Interventions to Achieve Early and Equitable Transplants (STEPS) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Northwell Health (Other); Geisinger Clinic (Other); University of Mississippi Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00097407; 7U01DK127918-02 (NIH); IHS-2020C1-19350-IC (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases
Keywords: Kidney transplant; Living donor kidney transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEPS Health System Surveillance and Outreach intervention (Experimental)
  Interventions: Behavioral: STEPS Health System Outreach intervention
- Usual Kidney Care (No Intervention)

INTERVENTIONS:
Behavioral: STEPS Health System Outreach intervention — STEPS Transplant Social Worker Education and Outreach, STEPS Transplant Coordinator Outreach
  Arms: STEPS Health System Surveillance and Outreach intervention

SUMMARY:
This project will study how kidney care for everyone despite race can reduce racial differences in care and improve access to kidney transplants, and specifically living donor kidney transplants (LDKT), for individuals with chronic kidney disease. A study focused on equality and patient needs (called 'STEPS') will 1) create a program to identify people who may need a kidney transplant ('STEPS Surveillance') and find people in health systems who may be able to receive kidney transplants early in their care and (2) study how well the 'STEPS Outreach' program works (comprised of transplant social workers and transplant coordinators who focus on equality and patient needs) compared to usual care to improve access to kidney transplants among Black and non-Black individuals as well as to improve access to transplants for everyone.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide oral informed consent
* Male or female, aged 18 to <=75 years
* Presence of CKD (2 eGFRs <60, 90 days apart) and at least 1 of the following: most recent eGFR less than 30 or KFRE greater than 10%
* English speaking with adequate ability to hear and understand questions over the phone
* Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Male or female, aged <18 or > 75 years
* Non-English speaking
* Lack of ability to hear and comprehend verbal communication.
* Patients on dialysis
* Deceased
* Hospice/palliative care
* Prior kidney transplant
* Currently waitlisted at any transplant center
* Self-reported terminal illness or receipt of hospice services

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1168 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Health system reported completion of transplant evaluation | 18 months
  Number of patients that said "yes" to the completion of transplant evaluation as reported in health system EHR and Administrative reports

SECONDARY OUTCOMES:
Live donor inquires to transplant center | 6 months, 12 months, 18 months
  the number of participants that made an inquiry to the transplant center related to live donors as reported in EHR or from questionnaire
Live kidney donor transplants | 6 months, 12 months, 18 months
  The number of participants that completed their live kidney donor transplant as reported by the EHR or questionnaire
Placement on deceased kidney donor waitlist | 6 months, 12 months, 18 months
  The number of patients that have been placed on the deceased kidney donor waitlist as reported in the EHR or UNOS
Deceased kidney donor transplants | 6 months, 12 months, 18 months
  The number of patients that received a deceased kidney donor transplant as reported in EHR or USRDS
Health system reported initiation of transplant evaluation | 18 months
  Number of patients that said "yes" to the initiation of transplant evaluation as reported in health system EHR and Administrative reports
Patient reported physician discussions | baseline, 6 months, 12 months, 18 months
  number of times patient talked to physician regarding kidney transplant measured by patient report in questionnaire
Patient reported family discussions | baseline, 6 months, 12 months, 18 months
  number of times patient talked to family regarding kidney transplant measured by patient reported in questionnaire
Patient reported initiation of transplant evaluation | baseline, 6 months, 12 months, 18 months
  Number of patients that said "yes" to the initiation of transplant evaluation measured by patient report in questionnaire
Patient reported completion of transplant evaluation | baseline, 6 months, 12 months, 18 months
  Number of patients that said "yes" to the completion of transplant evaluation measured by patient report in questionnaire
Patient reported identification of a living donor | baseline, 6 months, 12 months, 18 months
  Number of patients that said "yes" to the identification of a living donor measured by patient report in questionnaire
Patient reported kidney transplant knowledge | baseline, 6 months, 12 months, 18 months
  Number of questions patients correctly answer measured by patient report in questionnaire
Patient reported empowerment | baseline, 6 months, 12 months, 18 months
  Calculation of scaled questions from the adapted DES-SF form using a range of 1-5 for each question, with 5 being the best outcome, measured by patient report in questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ebony Boulware, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boulware LE, Ephraim PL, Shafi T, Green JA, Browne T, Strigo TS, Peskoe S, Wilson J, Lokhnygina Y, Alkon A, Jackson GL, Ellis MJ, Sudan D, Cameron B, Vaitla PK, Cabacungan A, Brubaker L, Obermiller EL, Diamantidis CJ. System Interventions to Achieve Early and Equitable Kidney Transplants (STEPS): Protocol for STEPS, a randomized comparative effectiveness clinical trial. Contemp Clin Trials. 2025 Jun;153:107911. doi: 10.1016/j.cct.2025.107911. Epub 2025 Apr 6. PMID 40199386

DOCUMENTS (1):
  • Informed Consent Form (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT05014256/ICF_000.pdf